CLINICAL TRIAL: NCT04792554
Title: Singapore Perioperative Ageing Study (Sing-PAS)
Status: Recruiting | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/00152
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Delirium; Aging; Myocardial Injury
Keywords: Geriatrics
MeSH Terms: conditions — Emergence Delirium | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Cohort: Elderly patients aged 65 and above who are planned for major non-cardiac surgery predicted to be at least 2 hours in duration and requiring at least 1 postoperative stay in hospital.
  Interventions: Other: Neurocognitive tests and blood taking

INTERVENTIONS:
Other: Neurocognitive tests and blood taking — Battery of neurocognitive tests and questionnaires including MoCA, PHQ-9, Falls History, FIFE, STOPBANG, Nutritional Survey, Global Physical Activity Questionnaire, Brief Pain Index, Brief Psychiatric Rating Scale, NuDESC, 3D-CAM. Blood taking.

SUMMARY:
The specific aim of the study will be to set up a perioperative database to longitudinally track the progress of elderly patients undergoing major surgery from the preoperative period to five years postoperatively. This database will form the foundation of a programme that will be sustainable through future grants to implement clinical strategies to improve outcomes.

DETAILED DESCRIPTION:
Singaporeans are rapidly ageing. One in every 4 Singaporeans will be aged 65 years and older in 2030, double the rate of that in 2015. Elderly patients have more chronic diseases and have a poorer recovery profile after illness or surgery. More recently, it has been reported that Singaporeans spend 10 years of their lives in poor health. Elderly patients are over-represented in patients coming for surgery, particularly for major cardiac and non-cardiac surgeries. While surgery is wonderful and lifesaving, the truth is that many elderly patients do not do well after major surgery. This was eloquently reported in the New York Times recently in an article titled "The Elderly Are Getting Complex Surgeries. Often It Doesn't End Well." Elderly patients value quality of life over quantity of life, but many are not aware of the long-term debilitation, organ dysfunction, pain, depression, economic burden and social strain that frequently accompanies major surgery. Elderly patients are more likely to lose independence after surgery, both physically and cognitively, and may never recover fully. There is clearly a disconnect between the elderly patient's (and their loved ones') expectations and reality. There is therefore a need to look closely at the operative journey of the elderly patient undergoing major surgery. Currently, clinical care is primarily concerned about achieving a technically successful surgery and recovery in the immediate postoperative phase, but there is much less oversight once the patient leaves the hospital system to community care. However, perioperative management significantly impacts the quality of life and activities of daily living for years after surgery. At NUHS, the MILES (Management and Innovation for Longevity in Elderly Surgical patients) programme has successfully reduced hospital length of stay of elderly patients undergoing abdominal surgery by addressing frailty and performing prehabilitation in selected patients. In this study, the study team intend to expand on this clinical programme to look at 3 primary concerns, namely postoperative delirium, trajectory of ageing, and myocardial injury, and the long-term implications of these concerns. Second, the team will incorporate biomarkers and other investigations to better risk profile patients, elucidate mechanistic processes, and provide better diagnostic and prognostic tools to clinicians. Third, the team will investigate the complimentary and detrimental roles of common systemic pathologies such as diabetes, anemia, renal dysfunction, malignancy, pain, and poor sleep on these outcomes. Therefore, the team intends to do a longitudinal study starting from the preoperative period up to 5 years after surgery in patients aged 65 years and above undergoing elective non-cardiac major surgery, defined as a surgery lasting at least 2 hours and requiring at least one day stay in hospital after surgery. It is envisioned that by using the data gained from this study, the investigators will be able to identify risk factors, trajectories of outcomes and gaps in their clinical care, and from there, formulate clinical strategies to address these gaps and mitigate the risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients aged 65 years and above
* Undergoing major non-cardiac surgery, defined as surgery that is predicted to be at least 2 hours and requiring at least 1 day postoperative stay in the hospital
* English, Chinese or Malay speaking
* Ability to provide informed consent

Exclusion Criteria:

* History of psychiatric disease
* Illiterate
* An active history of substance abuse.
* Undergoing neurological procedures
* Undergoing emergency surgeries
* Has a second surgery planned within 5 days of index surgery
* Non-resident of Singapore
* Severe hearing and/or speech impairment

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients aged 65 and above who are planned for major non-cardiac surgery predicted to be at least 2 hours in duration and requiring at least 1 postoperative stay in hospital.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Development of POD in elderly patients undergoing major non-cardiac surgery in a tertiary hospital in Singapore | Before surgery through to 5 years post surgery
  Collection of patient's demographics, medical records and surgical records to establish risk factors for POD development

CONTACTS AND LOCATIONS:
Overall Officials: Lian Kah Ti, Principal Investigator — National University Health System
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Alexandra Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rose J, Weiser TG, Hider P, Wilson L, Gruen RL, Bickler SW. Estimated need for surgery worldwide based on prevalence of diseases: a modelling strategy for the WHO Global Health Estimate. Lancet Glob Health. 2015 Apr 27;3 Suppl 2(Suppl 2):S13-20. doi: 10.1016/S2214-109X(15)70087-2. PMID 25926315
- [Background] Yang R, Wolfson M, Lewis MC. Unique Aspects of the Elderly Surgical Population: An Anesthesiologist's Perspective. Geriatr Orthop Surg Rehabil. 2011 Mar;2(2):56-64. doi: 10.1177/2151458510394606. PMID 23569671
- [Background] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Audisio R, Borozdina A, Cherubini A, Jones C, Kehlet H, MacLullich A, Radtke F, Riese F, Slooter AJ, Veyckemans F, Kramer S, Neuner B, Weiss B, Spies CD. European Society of Anaesthesiology evidence-based and consensus-based guideline on postoperative delirium. Eur J Anaesthesiol. 2017 Apr;34(4):192-214. doi: 10.1097/EJA.0000000000000594. PMID 28187050
- [Background] Evered L, Silbert B, Knopman DS, Scott DA, DeKosky ST, Rasmussen LS, Oh ES, Crosby G, Berger M, Eckenhoff RG; Nomenclature Consensus Working Group. Recommendations for the nomenclature of cognitive change associated with anaesthesia and surgery-2018. Br J Anaesth. 2018 Nov;121(5):1005-1012. doi: 10.1016/j.bja.2017.11.087. Epub 2018 Jun 15. PMID 30336844